CLINICAL TRIAL: NCT04696497
Title: Evaluation of Muscle Function at Discharge From ICU: Evaluation of the Correlation Between Manual Muscle Testing, Dynamometric and Peripheral Ultrasound Parameters
Brief Title: Muscle Function and Muscle Ultrasound in ICU
Acronym: DYNAMIQUE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulties and reorganization of the principal investigator's activity
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2020-02
Record Dates: First submitted 2020-12-04; First posted 2021-01-06 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Muscle Weakness
Keywords: Intensive care unit; Dynamometric; Ultrasound; Medical Research Council sum score; Ultrasonography; Muscle Strength; Critical Care
MeSH Terms: conditions — Muscle Weakness | interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscular Assessment (Other): All the patients will received the muscular assessments
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Dynamometric muscular assessment; Diagnostic Test: Manual muscular Assessment (MRC-SS)

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound measurements of muscle thickness, using a linear probe (high frequency) on four muscle groups:
  * Shoulder Side muscular compartment
  * Anterior Arm muscular compartment
  * Anterior thigh muscular compartment
  * Antero-lateral leg muscular compartment
Diagnostic Test: Dynamometric muscular assessment — The principle of electronic dynamometry is to measure an isometric force. To carry out these measurements, the examiner will stand on the side who has to be tested by exerting a pressure diametrically opposite to the patient's movement, thus preventing him/her from carrying out the movement. The patient will perform 3 tests for each movement, the best value will be collected by the examiner.
  The reference position is :
  Patient elbowed to the body bent at 90°, with trunk inclination at 30° in the resuscitation bed, lower limbs flat.
Diagnostic Test: Manual muscular Assessment (MRC-SS) — Following the same positions as for the dynamometer, the examiner will evaluate the 12 motor functions according to the following 60-point rating. With the maximum quote of 5 point representing normal strength and 0 point the total absence of any muscular contraction

SUMMARY:
The objective of intensive care therapists is to be able to detect as early as possible the muscle weakness acquired in intensive care, in order to implement curative strategies such as adapted nutrition and early rehabilitation. Various diagnostic tools are available for this purpose. To evaluate muscle mass, CT and MRI remain the gold standard but are difficult to implement in routine practice in ICU and are extremely expensive and can generate radiation for the patient.

Functional muscle evaluation is based on different voluntary tests which are not all able to predict muscle weakness acquired in ICU. In addition, some of the voluntary tests are expensive and require expert staff for practice and interpretation of results.

In addition, a muscle test such as MRC, although having an intraclass coefficient of 0.94, has little predictive value on clinical parameters such as mechanical ventilation duration and is not associated with mortality in the ward. However, it remains the test of choice to define a ICUAW with a threshold value of 48/60 points.

Dynamometry is a tool for measuring muscle strength. The patient is asked to perform a short and intense maximal muscular effort against manual or instrumental resistance. The limb segments must not move, it is an isometric effort. The most common measurement in intensive care units is the dynamometric grip force, called "handgrip".

In ICU, the patient may have touble with awareness, arousal or even comprehension, which will lead to biases in the evaluation of the motor force.

Ultrasound is a tool available in ICU and the muscle component can be assessed qualitatively or quantitatively without the patient's participation. Several studies have also demonstrated that muscle ultrasound is capable of reliably detecting pathological changes, particularly when repeated. Muscle ultrasound could thus help identify patients at higher risk of prolonged complications. Nevertheless, this technique lacks standardization and normative criteria (patient position, probe position, type and number of measurements, target muscle, etc.).

The main objective is to show that the dynamometric force relative to ultrasound thickness of several muscle groups (arm flexors/knee extensors/foot lifters) is correlated with manual MRC testing in intensive care unit (ICU) patients

DETAILED DESCRIPTION:
When the patient will be under invasive ventilatory support and coma, and will present the inclusion criteria, the investigator will perform ultrasound measurements of muscle thickness on four muscle groups:

* Shoulder Side muscular compartment
* Anterior Arm muscular compartment
* Anterior thigh muscular compartment
* Antero-lateral leg muscular compartment The ultrasound measurements will be made once a day each weekday, until the discharge from ICU.

Ultrasound measurements will be stopped if the patient's condition deteriorates and the ICU team chooses to limit active therapy.

If the patient condition get better, the investigator will perform the first volitional muscle function assessment, as soon as the patient Glasgow scale will score 15/15:

1. Medical Research Council sum score (MRC-ss)
2. Dynamometric strength assessment with the muscular groups used for the MRC-ss Then the volitional muscle assessment will be made once every 3 days, until patient discharges from ICU.

ELIGIBILITY:
Inclusion Criteria:

* Major patient > 18 years old
* Admission for more than 24 hours in the ICU ward
* Stay must be at least 72 hours

Exclusion Criteria:

* Person with a neuromuscular pathology
* Person presenting an osteoarticular contraindication to mobilization
* Amputee
* Person under guardianship or curatorship
* Person not affiliated to a social security system
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between force/thickness ratio and MRC testing. | Day 28
  To show that the dynamometric force relative to ultrasound thickness of several muscle groups (arm flexors/knee extensors/foot lifters) is correlated with manual MRC testing in intensive care medicine patients

SECONDARY OUTCOMES:
Modification in millimeters of ultrasound muscle thickness | Day 28
  Modification in millimeters of ultrasound muscle thickness
Change in force measured by dynamometry in patients with more than 2 evaluations | Day 28
  Change in force measured by dynamometry in patients with more than 2 evaluations
Medical Research Council sum-score (MRC-ss) | Day 28
  Following the same positions as for the dynamometer evaluation, the examiner will evaluate the 12 motor functions according to the following 60-point rating. With the maximum quote of 5 point representing normal strength and 0 point the total absence of any muscular contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FOSSAT, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

REFERENCES:
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Apr 24;370(17):1626-35. doi: 10.1056/NEJMra1209390. No abstract available. PMID 24758618
- [Background] Hermans G, Van den Berghe G. Clinical review: intensive care unit acquired weakness. Crit Care. 2015 Aug 5;19(1):274. doi: 10.1186/s13054-015-0993-7. PMID 26242743
- [Background] Cheung AM, Tansey CM, Tomlinson G, Diaz-Granados N, Matte A, Barr A, Mehta S, Mazer CD, Guest CB, Stewart TE, Al-Saidi F, Cooper AB, Cook D, Slutsky AS, Herridge MS. Two-year outcomes, health care use, and costs of survivors of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Sep 1;174(5):538-44. doi: 10.1164/rccm.200505-693OC. Epub 2006 Jun 8. PMID 16763220
- [Background] Cuthbertson BH, Roughton S, Jenkinson D, Maclennan G, Vale L. Quality of life in the five years after intensive care: a cohort study. Crit Care. 2010;14(1):R6. doi: 10.1186/cc8848. Epub 2010 Jan 20. PMID 20089197
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312